CLINICAL TRIAL: NCT05147272
Title: Phase 1 Study of the PKMYT1 Inhibitor RP-6306 in Combination With Gemcitabine for the Treatment of Advanced Solid Tumors (MAGNETIC Study)
Brief Title: Study of RP-6306 With Gemcitabine in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study
Sponsor: Debiopharm International SA (Industry)
Collaborators: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-6306-02
Record Dates: First submitted 2021-11-10; First posted 2021-12-07 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Adult Solid Tumor
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Dose Escalation (Experimental): Multiple dose levels of RP-6306 and gemcitabine
  Interventions: Drug: RP-6306 (oral PKMYT1 inhibitor)

INTERVENTIONS:
Drug: RP-6306 (oral PKMYT1 inhibitor) — RP-6306 in combination with gemcitabine
  Other Names: Gemcitabine (IV)

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of RP-6306 in combination gemcitabine, in patients with eligible advanced solid tumors, determine the maximum tolerated dose (MTD) of RP-6306 in combination with gemcitabine, identify a recommended phase 2 dose (RP2D) and preferred schedule, examine preliminary pharmacokinetics (PK) and assess anti-tumor activity.

DETAILED DESCRIPTION:
Phase 1, multi-center, open-label, dose-escalation study to:

* Evaluate the safety profile and MTD of RP-6306 with gemcitabine to establish the RP2D and schedule
* Characterize the PK and pharmacodynamics of RP-6306 with gemcitabine
* Assess preliminary anti-tumor activity associated with RP-6306 with gemcitabine

The Sponsor of the study has changed from 'Repare Therapeutics' to 'Debiopharm International SA' in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and ≥18 years-of-age at the time of informed consent.
* ECOG Performance status 0 or 1.
* Locally advanced or metastatic resistant or refractory solid tumors.
* Submission of available tumor tissue at screening or willingness to have a biopsy performed if safe and feasible.
* Measurable disease as per RECIST v1.1.
* Ability to swallow and retain oral medications.
* Acceptable hematologic and organ function at screening.
* Negative pregnancy test (serum) for women of childbearing potential (WOCBP) at Screening.
* Resolution of all toxicities of prior therapy or surgical procedures.
* Life expectancy ≥12 weeks after the start of the treatment

Exclusion Criteria:

* Chemotherapy or small molecule antineoplastic agent given within 21 days or <5 half- lives, whichever is shorter, prior to first dose of study drug.
* History or current condition, therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation for the full duration of the study treatment.
* Patients who are pregnant or breastfeeding.
* Known sensitivity to any of the ingredients of RP-6306 or gemcitabine.
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction or other reasons which, in the investigator's opinion, could compromise the participating patient's safety.
* Major surgery within 4 weeks prior to first dose of RP-6306 and gemcitabine.
* Uncontrolled, symptomatic brain metastases.
* Uncontrolled hypertension.
* Moderate or severe hepatic impairment
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - # 1018, Mayo Clinic, Phoenix, Arizona
  - # 1019, UCLA, Westwood Cancer Center, Los Angeles, California
  - # 1017, Mayo Clinic, Jacksonville, Florida
  - # 1022, Moffitt Cancer Center, Tampa, Florida
  - # 1023, START Midwest, Grand Rapids, Michigan
  - # 1016, Mayo Clinic, Rochester, Minnesota
  - # 1008, Columbia University, New York, New York
  - # 1004, Memorial Sloan Kettering Cancer Institute, New York, New York
  - # 1010, University of Pennsylvania, Philadelphia, Pennsylvania
- # 2001, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- # 3003, Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine: 40 mg QD oral (PO) lunresertib continuously daily in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine: 80 mg QD oral (PO) lunresertib continuously daily in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine: 40 mg QD oral (PO) lunresertib continuously daily in combination with 600 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine: 40 mg BID oral (PO) lunresertib continuously daily in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine: 40 mg BID oral (PO) lunresertib continuously daily in combination with 600 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine: 40 mg BID oral (PO) lunresertib continuously daily in combination with 400 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine: 120 mg QD oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine: 120 mg QD oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 600 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine: 40 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine: 60 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 600 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day: 60 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 400 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8: 80 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8: 80 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 600 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
- Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8: 120 mg BID oral (PO) lunresertib for the first 3 day per week ( 3 days on/4 days off) in combination with 800 mg/m2 intravenous (IV) gemcitabine given over 30 minutes on Day 1 and 8 of each 21-day treatment cycle
Period: Overall Study
Arm/Group | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8
Started | 1 | 7 | 4 | 4 | 10 | 8 | 5 | 5 | 4 | 4 | 6 | 4 | 3 | 2
Completed | 0 | 2 | 0 | 0 | 5 | 3 | 0 | 2 | 0 | 3 | 2 | 0 | 1 | 0
Not Completed | 1 | 5 | 4 | 4 | 5 | 5 | 5 | 3 | 4 | 1 | 4 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Total
Number analyzed (Participants) | 1 | 7 | 4 | 4 | 10 | 8 | 5 | 5 | 4 | 4 | 6 | 4 | 3 | 2 | 67
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 66 (0) | 59.1 (8.53) | 71.0 (4.69) | 61 (10.85) | 61.4 (12.58) | 62.1 (10.69) | 62.4 (10.64) | 58.6 (6.73) | 66.0 (10.86) | 65.3 (5.19) | 62.5 (10.72) | 54.8 (4.58) | 75.0 (0.71) | 67.5 (9.59) | 62.6 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 3 | 3 | 8 | 8 | 5 | 5 | 3 | 4 | 3 | 2 | 3 | 2 | 57
  Male | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 6 | 4 | 4 | 10 | 7 | 5 | 3 | 2 | 3 | 5 | 4 | 3 | 2 | 59
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With of Treatment-related Adverse Event Data Per CTCAE v5.0 Criteria to Determine Safety and Tolerability of RP-6306 in Combination With Gemcitabine.
Description: Incidence of grade 3 and above Treatment Related Emergent Adverse Events (TRAEs)
Time Frame: Start of treatment to 30 days post last dose. up to 1.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8
Number analyzed (Participants) | 1 | 7 | 4 | 4 | 10 | 8 | 5 | 5 | 4 | 4 | 6 | 4 | 3 | 2
Participants | 0 | 3 | 3 | 4 | 8 | 7 | 5 | 5 | 1 | 3 | 4 | 1 | 3 | 2

2. Primary Outcome: Number of Dose Limiting Toxicities, as Defined Per Protocol, That Occur During the First Cycle (21 Days) of Treatment at Each Dose Level
Description: Evaluation of dose-limiting toxicities (DLTs) at or below a frequency of 25%
Time Frame: During 21 days from the initiation of the study treatment (C1D1)
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8
Number analyzed (Participants) | 1 | 6 | 3 | 3 | 10 | 7 | 3 | 4 | 4 | 3 | 4 | 3 | 3 | 2
Participants | 0 | 2 | 2 | 2 | 4 | 4 | 2 | 3 | 0 | 1 | 2 | 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days post last dose up to 1.5 years
Arm/Group | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8
All-Cause Mortality (participants affected / at risk) | 1/1 | 5/7 | 3/4 | 4/4 | 2/10 | 3/8 | 4/5 | 1/5 | 3/4 | 1/4 | 2/6 | 2/4 | 1/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 3/7 | 2/4 | 1/4 | 5/10 | 3/8 | 1/5 | 1/5 | 2/4 | 2/4 | 2/6 | 2/4 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7 | 4/4 | 4/4 | 10/10 | 8/8 | 5/5 | 5/5 | 4/4 | 4/4 | 6/6 | 4/4 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine (N=1) | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine (N=7) | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine (N=4) | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine (N=4) | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine (N=10) | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine (N=8) | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine (N=5) | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine (N=5) | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine (N=4) | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine (N=4) | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day (N=6) | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 (N=4) | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 (N=3) | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Module 1a: 40 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine (N=1) | Module 1a: 80 mg QD Lunresertib Continue + 800 mg/m2 Gemcitabine (N=7) | Module 1a: 80 mg QD Lunresertib Continue + 600 mg/m2 Gemcitabine (N=4) | Module 1a: 40 mg BID Lunresertib Continue + 800 mg/m2 Gemcitabine (N=4) | Module 1a: 40 mg BID Lunresertib Continue + 600 mg/m2 Gemcitabine (N=10) | Module 1a: 40 mg BID Lunresertib Continue + 400 mg/m2 Gemcitabine (N=8) | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine (N=5) | Module 1b: 120 mg QD Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine (N=5) | Module 1b: 40 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine (N=4) | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine (N=4) | Module 1b: 60 mg BID Lunresertib 3 Days on/4 Days Off + 400 mg/m2 Gemcitabine Day (N=6) | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 (N=4) | Module 1b: 80 mg BID Lunresertib 3 Days on/4 Days Off + 600 mg/m2 Gemcitabine Day 1 and 8 (N=3) | Module 1b: 120 mg BID Lunresertib 3 Days on/4 Days Off + 800 mg/m2 Gemcitabine Day 1 and 8 (N=2)
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 2 | 5 | 5 | 5 | 3 | 0 | 3 | 2 | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3 | 5 | 4 | 2 | 1 | 2 | 3 | 1 | 3 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 4 | 3 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 0 | 0 | 1 | 3 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 2 | 0 | 5 | 5 | 4 | 5 | 3 | 3 | 4 | 3 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 2 | 2 | 4 | 3 | 1 | 2 | 0 | 3 | 4 | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 4 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 3 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 3 | 1 | 5 | 7 | 5 | 4 | 4 | 2 | 3 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 1 | 4 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 0
Chills (General disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood lactate dehydrogenase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 3 | 3 | 2 | 2 | 3 | 3 | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 2 | 0 | 3 | 0 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 3 | 3 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 3 | 1 | 1 | 2 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 3 | 0 | 3 | 1 | 2 | 3 | 2 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Module 1a and 1b was conducted. However, Module 1c and 1d were not conducted, and the study was terminated early by the sponsor/company

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT05147272/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT05147272/SAP_001.pdf